CLINICAL TRIAL: NCT01584479
Title: Periodontal Disease Prevention Study:A Retrospective Cohort Study to Assess the Effect of Genetics and Dental Preventive Care on Periodontal Disease
Brief Title: Periodontal Disease Prevention Study
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, William Giannobile, Principal Investigator, University of Michigan
Other Study IDs: HUM00037624
Record Dates: First submitted 2012-04-12; First posted 2012-04-25 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Periodontitis
Keywords: periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Low Risk Experimental Group: 1 visit - Low Risk
  ~1200 subjects
  - Low Risk Experimental Group = 1 visit intervention, no history of periodontitis, non-smoker, non-diabetic, IL-1 genotype (-)
- Low risk Control Group: 2 visits - Low Risk
  ~1200 subjects
  - Low risk Control Group = 2 visit intervention, no history of periodontitis, non-smoker, non-diabetic, IL-1 genotype (-)
- High Risk Experimental Group: 1 visit - High Risk
  ~800 subjects High Risk Experimental Group = 1 visit intervention, one or more of the following risk factors: history of periodontitis, smoker or diabetic, IL-1 genotype (+)
- High Risk Control Group: 2 visits - High Risk
  ~800 subjects High Risk Control Group = 2 visit intervention, one or more of the following risk factors: history of periodontitis, smoker or diabetic, IL-1 genotype (+)

SUMMARY:
This study is one component of a program to improve the maintenance of good dental health and the prevention of disease by use of risk stratification methods to efficiently guide increased preventive services to adult dental patients who are at increased risk for the major dental diseases, caries and adult periodontitis.

The investigators will use a retrospective cohort model to analyze a large dental claims database to determine if the frequency of preventive services influenced the periodontal disease outcomes and to determine if periodontal risk assessment information can be used to stratify dental patients into "high risk" and "low risk" categories that influence the effect of preventive services on periodontitis outcomes.

Primary Objective To evaluate whether dental patients who are classified as "low risk" for periodontal disease progression, based on history of periodontitis (claims history), smoking, diabetes, and IL-1 genetic variations, have different primary and secondary endpoints if they had two dental cleanings per year compared to one cleaning per year.

Secondary Objectives To evaluate whether dental patients who are classified as "high risk" for periodontal disease progression, based on a history of periodontitis, smoking, diabetes, and IL-1 genetic variations, have different primary and secondary endpoints if they had two dental cleanings per year compared to one cleaning per year.

To evaluate whether dental patients who have had one dental cleaning per year have different primary and secondary endpoints if they are classified as "low risk" for periodontal disease compared to patients who are classified as "high risk." To evaluate whether dental patients who have had two dental cleaning per year have different primary and secondary endpoints if they are classified as "low risk" for periodontal disease compared to patients who are classified as "high risk."

ELIGIBILITY:
Inclusion Criteria:

* Study may include all participants who are 34-55 years old in 1992 (48-68 years old in 2010) and who have at least a 15-year dental claim history with Delta Dental.

Exclusion Criteria:

* Organ transplant recipients are excluded.

Ages: 34 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study may include all participants who are 34-55 years old in 1992 (48-68 years old in 2010) and who have at least a 15-year dental claim history with Delta Dental.
Sampling Method: Probability Sample
Enrollment: 5117 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Giannobile, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Giannobile WV, Braun TM, Caplis AK, Doucette-Stamm L, Duff GW, Kornman KS. Patient stratification for preventive care in dentistry. J Dent Res. 2013 Aug;92(8):694-701. doi: 10.1177/0022034513492336. Epub 2013 Jun 10. PMID 23752171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 25,452 individuals meeting inclusion criteria, 9,927 (0.39 of eligible) consented to participate, and 5,117(0.515 of consented) returned completed questionnaires and were successfully genotyped.
Groups:
- Low Risk Experimental Group: 1 visit - Low Risk 732 evaluable subjects
  - Low Risk Experimental Group = 1 visit intervention, no history of periodontitis, non-smoker, non-diabetic, IL-1 genotype (-)
- Low Risk Control Group: 2 visits - Low Risk 1,668 evaluable subjects
  - Low risk Control Group = 2 visit intervention, no history of periodontitis, non-smoker, non-diabetic, IL-1 genotype (-)
- High Risk Experimental Group: 1 visit - High Risk 852 evaluable subjects
  High Risk Experimental Group = 1 visit intervention, one or more of the following risk factors: history of periodontitis, smoker or diabetic, IL-1 genotype (+)
- High Risk Control Group: 2 visits - High Risk 1,847 evaluable subjects
  High Risk Control Group = 2 visit intervention, one or more of the following risk factors: history of periodontitis, smoker or diabetic, IL-1 genotype (+)
Period: Overall Study
Arm/Group | Low Risk Experimental Group | Low Risk Control Group | High Risk Experimental Group | High Risk Control Group
Started | 732 | 1686 | 852 | 1847
Completed | 732 | 1686 | 852 | 1847
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: See Giannobile et al 2013 manuscript included
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Experimental Group | Low Risk Control Group | High Risk Experimental Group | High Risk Control Group | Total
Number analyzed (Participants) | 732 | 1686 | 852 | 1847 | 5117
Age, Customized [Number; unit: participants] — The participants analyzed had to be within this age range during the year 2010.
  participants
    >34 and < 55 years | 732 | 1686 | 852 | 1847 | 5117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 1130 | 537 | 1238 | 3366
  Male | 271 | 556 | 315 | 609 | 1751
Region of Enrollment [Number; unit: participants]
  United States | 732 | 1686 | 852 | 1847 | 5117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tooth Loss Over 16 Year Period
Description: Tooth loss rate over 16 years was calculated as the cumulative percentage of participants with tooth loss over 16 years.
Time Frame: 16 years
Measure: Number; unit: percentage of participants
Arm/Group | Low Risk Experimental Group | Low Risk Control Group | High Risk Experimental Group | High Risk Control Group
Number analyzed (Participants) | 732 | 1686 | 852 | 1847
percentage of participants | 16.4 | 13.8 | 22.1 | 16.9

2. Secondary Outcome: Change in Total Dental Claims During Monitoring Period
Time Frame: 10 and 15 years
Reporting Status: Not Posted

3. Secondary Outcome: Change in Total Periodontal Claims During the Monitoring Period
Time Frame: 10 and 15 years
Reporting Status: Not Posted

4. Secondary Outcome: Change in Periodontal Surgery Claims
Time Frame: 10 and 15 years
Reporting Status: Not Posted

5. Secondary Outcome: Change in Relationship of Risk Category & Tooth Loss Rate With Systemic Disease History on Questionnaire.
Time Frame: 10 and 15 years
Reporting Status: Not Posted

6. Secondary Outcome: Change in Evaluation for Dental Caries and Oral Cancer Within the Risk Categories
Time Frame: 10 and 15 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: This is an survey research study with the patient collection of their own biological specimen and the filling out of a survey to release their payer data (non-interventional).
Arm/Group | Low Risk Experimental Group | Low Risk Control Group | High Risk Experimental Group | High Risk Control Group
Serious Adverse Events (participants affected / at risk) | 0/732 | 0/1686 | 0/852 | 0/1847
Other Adverse Events (participants affected / at risk) | 0/732 | 0/1686 | 0/852 | 0/1847

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No